CLINICAL TRIAL: NCT00299494
Title: A Phase 1/2 Study Of Cmc-544 Administered In Combination With Rituximab In Subjects With Follicular Or Diffuse Large B-cell Non-hodgkin's Lymphoma
Brief Title: Study Evaluating Inotuzumab Ozogamicin [CMC-544] Administered In Combination With Rituximab In Subjects With Non-Hodgkin's Lymphoma (NHL)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 3129K3-101; B1931004 (Other: Alias Study Number); 2005-005436-27 (EudraCT Number)
Record Dates: First submitted 2006-03-02; First posted 2006-03-06 (Estimated); Results first posted 2018-03-08 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-02

CONDITIONS: B-Cell Lymphoma
Keywords: Lymphoma; NHL
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma | interventions — Inotuzumab Ozogamicin; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB (FOLLICULAR) (Experimental): Follicular
  Interventions: Drug: inotuzumab ozogamicin; Drug: Rituximab
- INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB (DLBCL) (Experimental): Diffuse Large B-cell Lymphoma
  Interventions: Drug: inotuzumab ozogamicin; Drug: Rituximab
- INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB (REFRACTORY) (Experimental): Refractory Aggressive NHL
  Interventions: Drug: inotuzumab ozogamicin; Drug: Rituximab

INTERVENTIONS:
Drug: inotuzumab ozogamicin — IV, 1.8 mg/m2, q4w
  Other Names: CMC-544
  Arms: INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB (FOLLICULAR)
Drug: inotuzumab ozogamicin — IV, 1.8 mg/m2, q4w
  Other Names: CMC-544
  Arms: INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB (DLBCL)
Drug: inotuzumab ozogamicin — IV, 1.8 mg/m2, q4w
  Other Names: CMC-544
  Arms: INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB (REFRACTORY)
Drug: Rituximab — rituximab 375 mg/m^2 via IV infusion on Day 1

SUMMARY:
The purpose of the study is to determine the tolerability, the initial safety profile and maximum tolerated dose, and to obtain preliminary information on the antitumor activity of inotuzumab ozogamicin [CMC-544] in combination with rituximab in subjects with follicular, diffuse large B-Cell, or mantle cell NHL.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with CD20 and CD22-positive, follicular or diffuse large B-cell NHL who have not responded or progressed after 1 or 2 prior therapies; or subjects with CD20 and CD22-positive intermediate/aggressive NHL (diffuse large B-cell, mantle cell, transformed follicular or follicular grade 3b NHL) who have not responded or progressed after 1 or more prior therapies and are refractory to a previous rituximab containing therapy.
* Prior therapy must contain at least one course of rituximab therapy, as single agent or in combination.
* Measurable disease.

Exclusion Criteria:

* Subjects who are candidates for other potentially curative therapies.
* Subjects must not have received previous radioimmunotherapy.
* Subjects who have undergone a prior bone marrow transplantation within the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2006-05-04 (Actual); Primary Completion 2014-05-19 (Actual); Study Completion 2014-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (37):
- United States (18):
  - University of Alabama at Birmingham-, Birmingham, Alabama
  - IDS Pharmacy, Birmingham, Alabama
  - California Cancer Care, Inc., Greenbrae, California
  - University of California Medical Center, San Francisco, California
  - California Cancer Care, San Mateo, California
  - Emory Clinic, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Emory University Investigational Drug Service, Atlanta, Georgia
  - Northwestern Medical Faculty Foundation, Chicago, Illinois
  - Nevada Cancer Institute-, Las Vegas, Nevada
  - Rosewell Park Cancer Institute, Buffalo, New York
  - Gabrail Cancer Center, Canton, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Gabrail Cancer Center, Dover, Ohio
  - UHHS - Westlake, Westlake, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
- Royal Brisbane and Women's Hospital, Herston, Brisbane, QLD, Australia
- Belgium (3):
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven, Vlaams-brabant
  - Universitair Ziekenhuis Gent, Ghent
  - University Hospital Gent - Department of Hematology, Ghent
- France (3):
  - Hôpital André MIGNOT, Le Chesnay
  - Hôpital Saint-Louis, Paris
  - CH Lyon Sud, Pierre-Bénite
- Germany (2):
  - Universitaetsklinik Bonn, Medizinische Klinik und Poliklinik III, Bonn
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet, III. medizinische klinik und Poliklinik, Mainz
- Prince Of Wales Hospital, Shatin N.T., HONG KONG, Hong Kong
- Universita La Sapienza Cattedra di Ematologia, Roma, Italy
- Erasmus Medisch Centrum--, Rotterdam, South Holland, Netherlands
- Centrum Onkologii-Instytut im. Marii Sklodowskiej-Curie, Warsaw, Poland
- Asan Medical Center, Seoul, South Korea
- Hospital Clinic I Provincial de Barcelona, Barcelona, Spain
- University Hospital Zurich, Zurich, Switzerland
- United Kingdom (3):
  - Derriford Hospital - Plymouth, Plymouth, Devon
  - Somers Cancer Science Building MP824, Southampton, Hampshire
  - Bart's Cancer Institute; Queen Mary University of London, London

REFERENCES:
- [Derived] Fayad L, Offner F, Smith MR, Verhoef G, Johnson P, Kaufman JL, Rohatiner A, Advani A, Foran J, Hess G, Coiffier B, Czuczman M, Gine E, Durrant S, Kneissl M, Luu KT, Hua SY, Boni J, Vandendries E, Dang NH. Safety and clinical activity of a combination therapy comprising two antibody-based targeting agents for the treatment of non-Hodgkin lymphoma: results of a phase I/II study evaluating the immunoconjugate inotuzumab ozogamicin with rituximab. J Clin Oncol. 2013 Feb 10;31(5):573-83. doi: 10.1200/JCO.2012.42.7211. Epub 2013 Jan 7. PMID 23295790
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3129K3-101&StudyName=Study%20Evaluating%20CMC-544%20Administered%20In%20Combination%20With%20Rituximab%20In%20Subjects%20With%20Non-Hodgkin%27s%20Lymphoma%20%28NHL%29

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A Open-Label, Phase 1/2 Study of CMC-544 (Inotuzumab Ozogamicin) in Combination With Rituximab in Subjects
Pre-assignment Details: Eligible Subjects were Randomly Assigned to Study Treatments
Groups:
- INOTUZUMAB OZOGAMICIN 0.8 MG/M^2 + RITUXIMAB 375 MG/M^2: Participants received rituximab 375 mg/m^2 via intravenous (IV) infusion on Day 1 and inotuzumab ozogamicin 0.8 mg/m^2 via IV infusion on Day 2 of each 28-day cycle for up to 8 cycles unless there was evidence of progressive disease, unacceptable toxicity, or the participant refused further treatment.
- INOTUZUMAB OZOGAMICIN 1.3 MG/M^2 + RITUXIMAB 375 MG/M^2: Participants received rituximab 375 mg/m^2 via IV infusion on Day 1 and inotuzumab ozogamicin 1.3 mg/m^2 via IV infusion on Day 2 of each 28-day cycle for up to 8 cycles unless there was evidence of progressive disease, unacceptable toxicity, or the participant refused further treatment.
- INOTUZUMAB OZOGAMICIN 1.8 MG/M^2 + RITUXIMAB 375 MG/M^2: Participants received rituximab 375 mg/m^2 via IV infusion on Day 1 and inotuzumab ozogamicin 1.8 mg/m^2 via IV infusion on Day 2 of each 28-day cycle for up to 8 cycles unless there was evidence of progressive disease, unacceptable toxicity, or the participant refused further treatment.
- INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (FOLLICULAR): Participants received the maximum tolerated dose (MTD) determined in the dose escalation phase; MTD determination in the dose escalation phase was based on toxicities during the 1st cycle. Participants with follicular lymphoma received rituximab 375 mg/m^2 via IV infusion on Day 1 and the MTD of inotuzumab ozogamicin (1.8 mg/m^2) via IV infusion on Day 2 of each 28-day cycle for up to 8 cycles unless there was evidence of progressive disease, unacceptable toxicity, or the participant refused further treatment.
- INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (DLBCL): Participants received the MTD determined in the dose escalation phase; MTD determination in the dose escalation phase was based on toxicities during the 1st cycle. Participants with diffuse large B-cell lymphoma (DLBCL) received rituximab 375 mg/m^2 via IV infusion on Day 1 and the MTD of inotuzumab ozogamicin (1.8 mg/m^2) via IV infusion on Day 2 of each 28-day cycle for up to 8 cycles unless there was evidence of progressive disease, unacceptable toxicity, or the participant refused further treatment.
- INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (REFRACTORY): Participants received the MTD determined in the dose escalation phase; MTD determination in the dose escalation phase was based on toxicities during the first cycle. Participants with either refractory aggressive or intermediate B-cell non-Hodgkin's lymphoma (NHL) received rituximab 375 mg/m^2 via IV infusion on Day 1 and the MTD of inotuzumab ozogamicin (1.8 mg/m^2) via IV infusion on Day 2 of each 28-day cycle for up to 8 cycles unless there was evidence of progressive disease, unacceptable toxicity, or the participant refused further treatment.
Period: Overall Study
Arm/Group | INOTUZUMAB OZOGAMICIN 0.8 MG/M^2 + RITUXIMAB 375 MG/M^2 | INOTUZUMAB OZOGAMICIN 1.3 MG/M^2 + RITUXIMAB 375 MG/M^2 | INOTUZUMAB OZOGAMICIN 1.8 MG/M^2 + RITUXIMAB 375 MG/M^2 | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (FOLLICULAR) | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (DLBCL) | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (REFRACTORY)
Started | 5 | 3 | 7 | 34 | 40 (1 participant received rituximab only, and did not receive inotuzumab ozogamicin) | 30
Completed | 2 | 2 | 3 | 24 | 13 | 4
Not Completed | 3 | 1 | 4 | 10 | 27 | 26
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 3 | 1 | 4
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Death | 3 | 1 | 4 | 6 | 18 | 19
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 3 | 1
Not completed — Other - Unspecified | 0 | 0 | 0 | 0 | 3 | 1
Not completed — Other - site closure | 0 | 0 | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population: All participants enrolled into the intended dose scheme.
Groups:
- INOTUZUMAB OZOGAMICIN 0.8 MG/M^2 + RITUXIMAB 375 MG/M^2: Participants received rituximab 375 mg/m^2 via IV infusion on Day 1 and inotuzumab ozogamicin 0.8 mg/m^2 via IV infusion on Day 2 of each 28-day cycle for up to 8 cycles unless there was evidence of progressive disease, unacceptable toxicity, or the participant refused further treatment.
- INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (FOLLICULAR): Participants received the MTD determined in the dose escalation phase; MTD determination in the dose escalation phase was based on toxicities during the 1st cycle. Participants with follicular lymphoma received rituximab 375 mg/m^2 via IV infusion on Day 1 and the MTD of inotuzumab ozogamicin (1.8 mg/m^2) via IV infusion on Day 2 of each 28-day cycle for up to 8 cycles unless there was evidence of progressive disease, unacceptable toxicity, or the participant refused further treatment.
- INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (DLBCL): Participants received the MTD determined in the dose escalation phase; MTD determination in the dose escalation phase was based on toxicities during the 1st cycle. Participants with DLBCL received rituximab 375 mg/m^2 via IV infusion on Day 1 and the MTD of inotuzumab ozogamicin (1.8 mg/m^2) via IV infusion on Day 2 of each 28-day cycle for up to 8 cycles unless there was evidence of progressive disease, unacceptable toxicity, or the participant refused further treatment.
- INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (REFRACTORY): Participants received the MTD determined in the dose escalation phase; MTD determination in the dose escalation phase was based on toxicities during the 1st cycle. Participants with either refractory aggressive or intermediate B-cell NHL received rituximab 375 mg/m^2 via IV infusion on Day 1 and the MTD of inotuzumab ozogamicin (1.8 mg/m^2) via IV infusion on Day 2 of each 28-day cycle for up to 8 cycles unless there was evidence of progressive disease, unacceptable toxicity, or the participant refused further treatment.
- Total: Total of all reporting groups
Arm/Group | INOTUZUMAB OZOGAMICIN 0.8 MG/M^2 + RITUXIMAB 375 MG/M^2 | INOTUZUMAB OZOGAMICIN 1.3 MG/M^2 + RITUXIMAB 375 MG/M^2 | INOTUZUMAB OZOGAMICIN 1.8 MG/M^2 + RITUXIMAB 375 MG/M^2 | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (FOLLICULAR) | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (DLBCL) | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (REFRACTORY) | Total
Number analyzed (Participants) | 5 | 3 | 7 | 34 | 40 | 30 | 119
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.4 (10.9) | 65.7 (0.6) | 60.7 (9.6) | 61.7 (12.2) | 67.2 (13.0) | 55.5 (15.8) | 62.1 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 18 | 17 | 9 | 48
  Male | 3 | 2 | 6 | 16 | 23 | 21 | 71

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Inotuzumab Ozogamicin in Combination With Rituximab (375 mg/m^2 )
Description: Inotuzumab ozogamicin was dose escalated (3 to 6 evaluable participants enrolled per dose cohort) during the first 28 days after the first administration of inotuzumab ozogamicin + rituximab. Enrollment at the next dose level or enrollment of additional subjects into a cohort proceeded according to the following criteria: 0 dose-limiting toxicity (DLT) by Day 28 of first dose move to higher dose, 1 participant reporting DLT but no others in cohort by Day 28 of first dose move to higher dose, greater than 2 participants reporting DLT by Day 28 of first dose stop and prior dose level considered MTD. The worldwide medical monitor and investigators reviewed all significant study drug-related toxicities to determine if the dose escalation rules were satisfied and whether the dose escalation schedule required modification.
Time Frame: First 28-day cycle
Population: Intent-To-Treat (ITT) Population: All participants included in the intended dose scheme. One additional participant was enrolled over the 6 planned participants in 1.8 mg/m^2 dose cohort because 1 participant was unevaluable for MTD evaluations.
Measure: Number; unit: mg/m^2
Groups:
- INOTUZUMAB OZOGAMICIN + RITUXIMAB 375 MG/M^2: Participants received rituximab 375 mg/m^2 via IV infusion on Day 1 and inotuzumab ozogamicin (0.8 mg/m^2, 1.3 mg/m^2, or 1.8 mg/m^2) via IV infusion on Day 2 of each 28-day cycle for up to 8 cycles unless there was evidence of progressive disease, unacceptable toxicity, or the participant refused further treatment.
Arm/Group | INOTUZUMAB OZOGAMICIN + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 15
mg/m^2 | 1.8

2. Primary Outcome: Percentage of Participants With a Treatment Emergent Adverse Event (TEAE) (Safety Population)
Description: A TEAE is any event that occurred after the first dose of study drug up to 56 days post the last dose of study drug (either rituximab or inotuzumab ozogamicin).
Time Frame: Protocol reporting period of from informed consent to at least 28 days after the last dose. This outcome measure time frame: From the first dose of study drug to up to 56 days after the last dose of either study drug.
Population: Safety population: All participants receiving at least 1 dose of inotuzumab ozogamicin or rituximab.
Measure: Number; unit: Percentage of participants
Arm/Group | INOTUZUMAB OZOGAMICIN 0.8 MG/M^2 + RITUXIMAB 375 MG/M^2 | INOTUZUMAB OZOGAMICIN 1.3 MG/M^2 + RITUXIMAB 375 MG/M^2 | INOTUZUMAB OZOGAMICIN 1.8 MG/M^2 + RITUXIMAB 375 MG/M^2 | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (FOLLICULAR) | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (DLBCL) | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (REFRACTORY)
Number analyzed (Participants) | 5 | 3 | 7 | 34 | 40 | 30
Percentage of participants
  % participants with a TEAE | 100 | 100 | 100 | 100 | 100 | 100
  % participants with serious TEAE | 20.0 | 0 | 14.3 | 26.5 | 30.0 | 16.7
  % participants with Grade 3 or 4 TEAE | 80.0 | 66.7 | 71.4 | 67.6 | 75.0 | 63.3
  % participants with Grade 5 TEAE | 20.0 | 0 | 0 | 0 | 2.5 | 6.7
  % participants for study drug discontinuation | 0 | 33.3 | 28.6 | 61.8 | 50.0 | 33.3
  % participants with dose reduction due to TEAE | 0 | 0 | 14.3 | 14.7 | 10.0 | 0
  % participants for study drug stopped temporarily | 20.0 | 0 | 42.9 | 44.1 | 40.0 | 10.0

3. Secondary Outcome: Percentage of Participants With Complete Response (CR), Unconfirmed CR (CRu), or Partial Response (PR)
Description: CR: a. Complete disappearance of all detectable clinical and radiographic evidence of disease, disease-related symptoms, and normalization of NHL assignable biochemical abnormalities ; b. lymph nodes and nodal masses must have regressed to normal size; c. Spleen regressed in size and not palpable on physical exam, size of other organs enlarged due to disease decreased in size; d. Repeat bone marrow infiltrate clear. CRu: CR but allows for a. Residual lymph node mass >1.5 cm in greatest transverse diameter has regressed by more than 75% in diameter. Individual nodes that were previously confluent regressed more than 75 % in their product diameters; b. Indeterminate bone marrow. PR: a. ≥50 % decrease in product of the diameters (SPD) of the 6 largest dominant nodes or nodal masses; b. No increase in size of other nodes, liver, or spleen, c. Liver or spleen nodules regressed ≥50% in the SPD; d. Other organs usually assessable, no measurable disease present.
Time Frame: Approximately every 2 (during treatment) or 3 (during follow-up) to 6 months for up to 5 years from 1st dose
Population: ITT population: all participants enrolled into the intended dose scheme. Using exact method based on binomial distribution.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | INOTUZUMAB OZOGAMICIN 0.8 MG/M^2 + RITUXIMAB 375 MG/M^2 | INOTUZUMAB OZOGAMICIN 1.3 MG/M^2 + RITUXIMAB 375 MG/M^2 | INOTUZUMAB OZOGAMICIN 1.8 MG/M^2 + RITUXIMAB 375 MG/M^2 | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (FOLLICULAR) | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (DLBCL) | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (REFRACTORY)
Number analyzed (Participants) | 5 | 3 | 7 | 34 | 40 | 30
Percentage of participants | 40 [5.3 to 85.3] | 100 [29.2 to 100] | 57.1 [18.4 to 90.1] | 94.1 [80.3 to 99.3] | 72.5 [56.1 to 85.4] | 20 [7.7 to 38.6]

4. Secondary Outcome: Kaplan-Meier Estimates of Progression Free Survival (PFS)
Description: The Kaplan-Meier method was used to determine PFS. 95% 2-sided confidence interval were calculated using stratified Cox proportional hazard regression. Relapsed or Progressive Disease (PD) requires the following: a. Appearance of any new lesions, b. Increase by >= 50% in the size of previously involved sites, c. >= 50% increase in greatest diameter of any previously identified node greater than 1 cm in its short axis or in the SPD of more than one node, d. >= 50% increase from nadir in the product diameter of any previously identified abnormal node for PRs or nonresponders, e. Enlarging spleen or liver.
Time Frame: From the date of first dose of test article until the first date on which disease progression or death was documented or new anticancer start, any of which could be reported up to 5 years post last dose
Population: ITT population. Calculated using Kaplan-Meier method.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | INOTUZUMAB OZOGAMICIN 0.8 MG/M^2 + RITUXIMAB 375 MG/M^2 | INOTUZUMAB OZOGAMICIN 1.3 MG/M^2 + RITUXIMAB 375 MG/M^2 | INOTUZUMAB OZOGAMICIN 1.8 MG/M^2 + RITUXIMAB 375 MG/M^2 | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (FOLLICULAR) | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (DLBCL) | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (REFRACTORY)
Number analyzed (Participants) | 5 | 3 | 7 | 34 | 40 | 30
Months | 1.7 [0.3 to NA] — insufficient data to calculate | NA [21.2 to NA] — insufficient data to calculate | NA [1.7 to NA] — insufficient data to calculate | NA [NA to NA] — insufficient data to calculate | 17.1 [6.8 to 56.6] | 1.8 [1.0 to 3.9]

5. Secondary Outcome: Kaplan-Meier Estimates of the Probability of Being Progression Free at 6 Months
Description: Progression Free Survival is defined as the time interval from the first dose of test article until the first date on which relapsed disease, progression, initiation of new anti-cancer treatment due to persistent/refractory disease, or death was documented, censored at the last tumor evaluation.
Time Frame: From the first dose to 6 months after first dose
Population: ITT population; Calculated using Kaplan-Meier method.
Measure: Number (95% Confidence Interval); unit: Probability
Groups:
- INOTUZUMAB OZOGAMICIN 0.8 MG/M^2: Participants received rituximab 375 mg/m^2 via IV infusion on Day 1 and inotuzumab ozogamicin 0.8 mg/m^2 via IV infusion on Day 2 of each 28-day cycle for up to 8 cycles unless there was evidence of progressive disease, unacceptable toxicity, or the participant refused further treatment.
Arm/Group | INOTUZUMAB OZOGAMICIN 0.8 MG/M^2 | INOTUZUMAB OZOGAMICIN 1.3 MG/M^2 + RITUXIMAB 375 MG/M^2 | INOTUZUMAB OZOGAMICIN 1.8 MG/M^2 + RITUXIMAB 375 MG/M^2 | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (FOLLICULAR) | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (DLBCL) | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (REFRACTORY)
Number analyzed (Participants) | 5 | 3 | 7 | 34 | 40 | 30
Probability | 0.4 [0.1 to 0.8] | 1.0 [NA to NA] — Insufficient data to calculate | 0.6 [0.2 to 0.8] | 1.0 [NA to NA] — Insufficient data to calculate | 0.7 [0.5 to 0.8] | 0.2 [0.1 to 0.4]

6. Secondary Outcome: Kaplan-Meier Estimates of Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause, censoring at the date of last contact. The Kaplan-Meier method was used to determine OS. 95% 2-sided confidence interval were calculated using stratified Cox proportional hazard regression.
Time Frame: From the first dose up to 5 years post last dose
Population: ITT population. Calculated using Kaplan-Meier method.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | INOTUZUMAB OZOGAMICIN 0.8 MG/M^2 + RITUXIMAB 375 MG/M^2 | INOTUZUMAB OZOGAMICIN 1.3 MG/M^2 + RITUXIMAB 375 MG/M^2 | INOTUZUMAB OZOGAMICIN 1.8 MG/M^2 + RITUXIMAB 375 MG/M^2 | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (FOLLICULAR) | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (DLBCL) | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (REFRACTORY)
Number analyzed (Participants) | 5 | 3 | 7 | 34 | 40 | 30
Months | 7.4 [0.5 to NA] — insufficient data to calculate | NA [21.7 to NA] — insufficient data to calculate | 16.9 [5.3 to NA] — insufficient data to calculate | NA [NA to NA] — insufficient data to calculate | 58.3 [34.8 to NA] — insufficient data to calculate | 8.4 [3.7 to 40.4]

7. Secondary Outcome: Kaplan-Meier Estimates of the Probability of Survival at 6 Months
Description: Overall Survival (OS) was defined as the time from randomization to death due to any cause, censoring at the date of last contact. The Kaplan-Meier method was used to determine OS. 95% 2-sided confidence interval were calculated using stratified Cox proportional hazard regression.
Time Frame: From the first dose to 6 months after first dose.
Population: ITT population. Calculated using Kaplan-Meier method.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | INOTUZUMAB OZOGAMICIN 0.8 MG/M^2 + RITUXIMAB 375 MG/M^2 | INOTUZUMAB OZOGAMICIN 1.3 MG/M^2 + RITUXIMAB 375 MG/M^2 | INOTUZUMAB OZOGAMICIN 1.8 MG/M^2 + RITUXIMAB 375 MG/M^2 | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (FOLLICULAR) | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (DLBCL) | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (REFRACTORY)
Number analyzed (Participants) | 5 | 3 | 7 | 34 | 40 | 30
Probability | 0.6 [0.1 to 0.9] | 1.0 [NA to NA] — insufficient data to calculate | 0.7 [0.3 to 0.9] | 1.0 [NA to NA] — insufficient data to calculate | 0.9 [0.8 to 1.0] | 0.6 [0.4 to 0.7]

8. Secondary Outcome: Kaplan-Meier Estimates of Time to Tumor Progression (TTP)
Description: TTP is defined as the interval from the first dose of the test article until the first date on which relapsed disease or progression, or death secondary to progression is documented, censored at the last disease assessment. Relapsed or Progressive Disease (PD) requires the following: a. Appearance of any new lesions, b. Increase by >= 50% in the size of previously involved sites, c. >= 50% increase in greatest diameter of any previously identified node greater than 1 cm in its short axis or in the SPD of more than one node, d. >= 50% increase from nadir in the product diameter of any previously identified abnormal node for PRs or nonresponders, e. Enlarging spleen or liver. The Kaplan-Meier method was used to determine TTP. 95% 2-sided confidence interval were calculated using stratified Cox proportional hazard regression.
Time Frame: From the date of first dose of test article until the first date on which disease progression or death was documented, any of which could be reported up to 5 years post last dose.
Population: ITT population. Calculated using Kaplan-Meier method.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- INOTUZUMAB OZOGAMICIN 0.8 MG/M^2 + RITUXIMAB 375 MG/M^2: Participants received rituximab 375 mg/m^2 via IV infusion on Day 1 and inotuzumab ozogamicin 0.8 mg/m^2 via IV infusion on Day 2 of each 28-day cycle for up to 8 cycles unless there was evidence of progressive disease, unacceptable toxicity, or the subject refused further treatment.
- INOTUZUMAB OZOGAMICIN 1.3 MG/M^2 + RITUXIMAB 375 MG/M^2: Participants received rituximab 375 mg/m^2 via IV infusion on Day 1 and inotuzumab ozogamicin 1.3 mg/m^2 via IV infusion on Day 2 of each 28-day cycle for up to 8 cycles unless there was evidence of progressive disease, unacceptable toxicity, or the subject refused further treatment.
- INOTUZUMAB OZOGAMICIN 1.8 MG/M^2 + RITUXIMAB 375 MG/M^2: Participants received rituximab 375 mg/m^2 via IV infusion on Day 1 and inotuzumab ozogamicin 1.8 mg/m^2 via IV infusion on Day 2 of each 28-day cycle for up to 8 cycles unless there was evidence of progressive disease, unacceptable toxicity, or the subject refused further treatment.
- INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (FOLLICULAR): Participants received the MTD determined in the dose escalation phase; MTD determination in the dose escalation phase was based on toxicities during the 1st cycle. Participants with follicular lymphoma received rituximab 375 mg/m^2 via IV infusion on Day 1 and the MTD of inotuzumab ozogamicin (1.8 mg/m^2) via IV infusion on Day 2 of each 28-day cycle for up to 8 cycles unless there was evidence of progressive disease, unacceptable toxicity, or the subject refused further treatment.
- INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (DLBCL): Participants received the MTD determined in the dose escalation phase; MTD determination in the dose escalation phase was based on toxicities during the 1st cycle. Participants with DLBCL received rituximab 375 mg/m^2 via IV infusion on Day 1 and the MTD of inotuzumab ozogamicin (1.8 mg/m^2) via IV infusion on Day 2 of each 28-day cycle for up to 8 cycles unless there was evidence of progressive disease, unacceptable toxicity, or the subject refused further treatment.
- INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (REFRACTORY): Participants received the MTD determined in the dose escalation phase; MTD determination in the dose escalation phase was based on toxicities during the 1st cycle. Participants with either refractory aggressive or intermediate B-cell NHL received rituximab 375 mg/m^2 via IV infusion on Day 1 and the MTD of inotuzumab ozogamicin (1.8 mg/m^2) via IV infusion on Day 2 of each 28-day cycle for up to 8 cycles unless there was evidence of progressive disease, unacceptable toxicity, or the subject refused further treatment.
Arm/Group | INOTUZUMAB OZOGAMICIN 0.8 MG/M^2 + RITUXIMAB 375 MG/M^2 | INOTUZUMAB OZOGAMICIN 1.3 MG/M^2 + RITUXIMAB 375 MG/M^2 | INOTUZUMAB OZOGAMICIN 1.8 MG/M^2 + RITUXIMAB 375 MG/M^2 | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (FOLLICULAR) | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (DLBCL) | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (REFRACTORY)
Number analyzed (Participants) | 5 | 3 | 7 | 34 | 40 | 30
Months | 1.7 [0.3 to NA] — insufficient data to calculate | NA [21.2 to NA] — insufficient data to calculate | NA [1.7 to NA] — insufficient data to calculate | NA [NA to NA] — insufficient data to calculate | 45.1 [15.2 to NA] — insufficient data to calculate | 1.7 [1.0 to 5.1]

9. Secondary Outcome: Kaplan-Meier Estimates of the Probability of Being Event Free at 6 Months
Description: Time-to-Tumor Progression (TTP): is defined as the interval from the first dose of the test article until the first date on which relapsed disease or progression, or death secondary to progression is documented, censored at the last disease assessment. Relapsed or Progressive Disease (PD) requires the following: a. Appearance of any new lesions, b. Increase by >=50% in the size of previously involved sites, c. >= 50% increase in greatest diameter of any previously identified node greater than 1 cm in its short axis or in the SPD of more than one node, d. >= 50% increase from nadir in the product diameter of any previously identified abnormal node for PRs or nonresponders, e. Enlarging spleen or liver. The Kaplan-Meier method was used to determineTTP. 95% 2-sided confidence interval were calculated using stratified Cox proportional hazard regression.
Time Frame: From enrollment to up to 6 months from 1st dose.
Population: ITT population. Calculated using Kaplan-Meier method.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | INOTUZUMAB OZOGAMICIN 0.8 MG/M^2 + RITUXIMAB 375 MG/M^2 | INOTUZUMAB OZOGAMICIN 1.3 MG/M^2 + RITUXIMAB 375 MG/M^2 | INOTUZUMAB OZOGAMICIN 1.8 MG/M^2 + RITUXIMAB 375 MG/M^2 | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (FOLLICULAR) | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (DLBCL) | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (REFRACTORY)
Number analyzed (Participants) | 5 | 3 | 7 | 34 | 40 | 30
Probability | 0.4 [0.1 to 0.8] | 1.0 [NA to NA] — insufficient data to calculate | 0.7 [0.3 to 0.9] | 1.0 [NA to NA] — insufficient data to calculate | 0.7 [0.5 to 0.9] | 0.3 [0.1 to 0.4]

10. Secondary Outcome: Duration of Response (CR+CRu+PR)
Description: Time from date measurement criteria met for CR, CRu, or PR (whichever occurred first) until first date relapsed disease/date of death. CR: Complete disappearance of all detectable clinical, radiographic evidence of disease, disease-related symptoms, normalization of NHL assignable biochemical abnormalities; lymph nodes, nodal masses regressed to normal size; spleen size regressed, not palpable on physical exam, size of other organs enlarged due to disease. CRu: CR but allows for: residual lymph node mass >1.5 cm in greatest transverse diameter that regressed >75% in product diameter. Individual nodes previously confluent, regressed by >75% in their product diameters; Indeterminate bone marrow. PR: ≥50% decrease in SPD of 6 largest dominant nodes/nodal masses; No increase in size of other nodes, liver, or spleen; Splenic/hepatic nodules regressed by ≥50% in SPD; Except splenic/hepatic nodules, involvement of other organs assessable and no measurable disease present.
Time Frame: Time from date measurement criteria are met for CR, CRu, or PR (whichever status is recorded first) until the first date relapsed disease or date of death (whichever occurs first) is objectively documented.
Population: ITT population. Calculated using Kaplan-Meier method using the number of participants that responded.
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | INOTUZUMAB OZOGAMICIN 0.8 MG/M^2 + RITUXIMAB 375 MG/M^2 | INOTUZUMAB OZOGAMICIN 1.3 MG/M^2 + RITUXIMAB 375 MG/M^2 | INOTUZUMAB OZOGAMICIN 1.8 MG/M^2 + RITUXIMAB 375 MG/M^2 | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (FOLLICULAR) | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (DLBCL) | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2 (REFRACTORY)
Number analyzed (Participants) | 5 | 3 | 7 | 34 | 40 | 30
Month | NA [14.4 to NA] — insufficient data to calculate | NA [17.7 to NA] — insufficient data to calculate | NA [3.0 to NA] — insufficient data to calculate | NA [NA to NA] — insufficient data to calculate | 43.2 [16.4 to NA] — insufficient data to calculate | 3.9 [2.3 to NA] — insufficient data to calculate

11. Secondary Outcome: Area Under the Serum Concentration-time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) of Inotuzumab Ozogamicin in Participants Receiving Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 on Dosing Day 30 and Day 58
Description: Serum concentration of inotuzumab ozogamicin on Dosing Days 30 and 58 were measured. AUCinf of inotuzumab ozogamicin was reported. AUCinf: AUClast (area under the serum concentration-time profile for inotuzumab ozogamicin from time zero to the time of the last quantifiable concentration) +(Clast [last quantifiable concentration]/kel [elimination rate constant]) where Clast is the predicted serum concentration of inotuzumab ozogamicin at the last quantifiable timepoint estimated from the log-linear regression analysis. Study Days Cycle 2, Days 30 (0, 1, 4 hours), 32, 36, 38, 43, 50, and 57 and Cycle 3, Days 58 (0, 1, 4 hours), 60, 64, 66, 71, 78, and 85 correspond to Dosing Day 30 for Cycle 2 and Dosing Day 58 for Cycle 3.
Time Frame: Cycle 2, Days 30 (0, 1, 4 hours), 32, 36, 38, 43, 50, and 57; Cycle 3, Days 58 (0, 1, 4 hours), 60, 64, 66, 71, 78, and 85
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.hr/mL
Groups:
- INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2: Participants received the MTD determined in the dose escalation phase; MTD determination in the dose escalation phase was based on toxicities during the 1st cycle. Participants with follicular lymphoma, DLBCL, and refractory aggressive or intermediate B-cell NHL received rituximab 375 mg/m^2 via IV infusion on Day 1 and the MTD of inotuzumab ozogamicin (1.8 mg/m^2) via IV infusion on Day 2 of each 28-day cycle for up to 8 cycles unless there was evidence of progressive disease, unacceptable toxicity, or the subject refused further treatment.
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
ng.hr/mL
  Dosing Day 30: number analyzed (Participants) | 32
  Dosing Day 30 | 36030 (34)
  Dosing Day 58: number analyzed (Participants) | 36
  Dosing Day 58 | 40550 (28)

12. Secondary Outcome: AUClast of Inotuzumab Ozogamicin in Participants Receiving Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 on Dosing Day 1, Day 30 and Day 58
Description: Serum concentration of inotuzumab ozogamicin on Dosing Days 1, 30 and 58 were measured. AUC of inotuzumab ozogamicin was reported. AUClast is area under the serum concentration-time profile from time zero to the time of the Clast, using Linear/Log trapezoidal method. Study Days Cycle 1, Days 1 (0 hour), 2 (0, 1, 4 hours), 4, 8, 10, 15, and 29; Cycle 2, Days 30 (0, 1, 4 hours), 32, 36, 38, 43, 50, and 57; and Cycle 3, Days 58 (0, 1, 4 hours), 60, 64, 66, 71, 78, and 85 correspond to Dosing Day 1 for Cycle 1; Dosing Day 30 for Cycle 2; and Dosing Day 58 for Cycle 3.
Time Frame: Cycle 1, Days 1 (0 hour), 2 (0, 1, 4 hours), 4, 8, 10, 15, and 29; Cycle 2, Days 30 (0, 1, 4 hours), 32, 36, 38, 43, 50, and 57; Cycle 3, Days 58 (0, 1, 4 hours), 60, 64, 66, 71, 78, and 85
Population: PK population: all participants dosed with inotuzumab ozogamicin.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
ng*h/mL
  Dosing Day 1: number analyzed (Participants) | 99
  Dosing Day 1 | 6157 (190)
  Dosing Day 30: number analyzed (Participants) | 86
  Dosing Day 30 | 9664 (76191)
  Dosing Day 58: number analyzed (Participants) | 71
  Dosing Day 58 | 17320 (225)

13. Secondary Outcome: Time of the Last Quantifiable Serum Concentration in a Dosing Interval (Tlast) of Inotuzumab Ozogamicin in Participants Receving Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 on Dosing Day 1, Day 30 and Day 58
Description: Tlast of inotuzumab ozogamicin on Dosing Days 1, 30, and 58 was reported. Tlast: Time of last quantifiable concentration of inotuzumab ozogamicin. Observed directly from data. Study Days Cycle 1, Days 1 (0 hour), 2 (0, 1, 4 hours), 4, 8, 10, 15, and 29; Cycle 2, Days 30 (0, 1, 4 hours), 32, 36, 38, 43, 50, and 57; and Cycle 3, Days 58 (0, 1, 4 hours), 60, 64, 66, 71, 78, and 85 correspond to Dosing Day 1 for Cycle 1; Dosing Day 30 for Cycle 2; and Dosing Day 58 for Cycle 3.
Time Frame: as for outcome 12
Population: PK population
Measure: Median (Full Range); unit: hr
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
hr
  Dosing Day 1: number analyzed (Participants) | 99
  Dosing Day 1 | 44.2 [1.00 to 192]
  Dosing Day 30: number analyzed (Participants) | 85
  Dosing Day 30 | 53.9 [4.00 to 647]
  Dosing Day 58: number analyzed (Participants) | 71
  Dosing Day 58 | 137 [1.00 to 647]

14. Secondary Outcome: Area Under the Steady-state Serum Concentration-time Curve (AUCtau) of Inotuzumab Ozogamicin in Participants Receving Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 on Dosing Day 1, Day 30 and Day 58
Description: Steady-state serum concentrations of inotuzumab ozogamicin on Dosing Days 1, 30 and 58 were measured. AUCtau of inotuzumab ozogamicin was reported. AUCtau=AUC over dosage interval tau calculated using Linear/log trapezoidal method. Study Days Cycle 1, Days 1 (0 hour), 2 (0, 1, 4 hours), 4, 8, 10, 15, and 29; Cycle 2, Days 30 (0, 1, 4 hours), 32, 36, 38, 43, 50, and 57; and Cycle 3, Days 58 (0, 1, 4 hours), 60, 64, 66, 71, 78, and 85 correspond to Dosing Day 1 for Cycle 1; Dosing Day 30 for Cycle 2; and Dosing Day 58 for Cycle 3.
Time Frame: as for outcome 12
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.hr/mL
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
ng.hr/mL
  Dosing Day 1: number analyzed (Participants) | 33
  Dosing Day 1 | 18660 (36)
  Dosing Day 30: number analyzed (Participants) | 32
  Dosing Day 30 | 35900 (28)
  Dosing Day 58: number analyzed (Participants) | 36
  Dosing Day 58 | 38820 (30)

15. Secondary Outcome: Peak Serum Concentration (Cmax) of Inotuzumab Ozogamicin in Participants Receving Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 on Dosing Day 1, Day 30 and Day 58
Description: Serum concentration of inotuzumab ozogamicin on Dosing Days 1, 30, and 58 were measured. Cmax of inotuzumab ozogamicin was reported. Cmax was observed directly from data. Study Days Cycle 1, Days 1 (0 hour), 2 (0, 1, 4 hours), 4, 8, 10, 15, and 29; Cycle 2, Days 30 (0, 1, 4 hours), 32, 36, 38, 43, 50, and 57; and Cycle 3, Days 58 (0, 1, 4 hours), 60, 64, 66, 71, 78, and 85 correspond to Dosing Day 1 for Cycle 1; Dosing Day 30 for Cycle 2; and Dosing Day 58 for Cycle 3.
Time Frame: as for outcome 12
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
ng/mL
  Dosing Day 1: number analyzed (Participants) | 101
  Dosing Day 1 | 600.2 (42)
  Dosing Day 30: number analyzed (Participants) | 89
  Dosing Day 30 | 378.3 (6435)
  Dosing Day 58: number analyzed (Participants) | 73
  Dosing Day 58 | 519.2 (586)

16. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) of Inotuzumab Ozogamicin in Participants Receiving Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 on Dosing Day 1, Day 30 and Day 58
Description: Tmax: Time at which Cmax occurs. Observed directly from data as time of first occurrence. Study Days Cycle 1, Days 1 (0 hour), 2 (0, 1, 4 hours), 4, 8, 10, 15, and 29; Cycle 2, Days 30 (0, 1, 4 hours), 32, 36, 38, 43, 50, and 57; and Cycle 3, Days 58 (0, 1, 4 hours), 60, 64, 66, 71, 78, and 85 correspond to Dosing Day 1 for Cycle 1; Dosing Day 30 for Cycle 2; and Dosing Day 58 for Cycle 3.
Time Frame: as for outcome 12
Population: PK population
Measure: Median (Full Range); unit: hr
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
hr
  Dosing Day 1: number analyzed (Participants) | 101
  Dosing Day 1 | 1.00 [0 to 192]
  Dosing Day 30: number analyzed (Participants) | 86
  Dosing Day 30 | 1.08 [0.583 to 479]
  Dosing Day 58: number analyzed (Participants) | 72
  Dosing Day 58 | 1.08 [0 to 647]

17. Secondary Outcome: Average Serum Concentration at Steady State (Cav) of Inotuzumab Ozogamicin in Participants Receiving Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 on Dosing Day 30 and Day 58
Description: Cav: AUCtau (Area under the concentration time profile)/tau for Dosing Day 30 Cycle 2 and Dosing Day 58 Cycle 3. Study Days Cycle 2, Days 30 (0, 1, 4 hours), 32, 36, 38, 43, 50, and 57 and Cycle 3, Days 58 (0, 1, 4 hours), 60, 64, 66, 71, 78, and 85 correspond to Dosing Day 30 for Cycle 2 and Dosing Day 58 for Cycle 3.
Time Frame: as for outcome 11
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
ng/mL
  Dosing Day 30: number analyzed (Participants) | 32
  Dosing Day 30 | 53.43 (28)
  Dosing Day 58: number analyzed (Participants) | 36
  Dosing Day 58 | 57.77 (30)

18. Secondary Outcome: Minimum Observed Serum Trough Concentration (Cmin) of Inotuzumab Ozogamicin in Participants Receiving Inotuzumab+Rituximab on Dosing Day 30 and Day 58
Description: Cmin: Lowest concentration observed during the dosing interval tau. Observed directly from data from Dosing Day 30 for Cycle 2; and Dosing Day 58 for Cycle 3. Study Days Cycle 2, Days 30 (0, 1, 4 hours), 32, 36, 38, 43, 50, and 57 and Cycle 3, Days 58 (0, 1, 4 hours), 60, 64, 66, 71, 78, and 85 correspond to Dosing Day 30 for Cycle 2 and Dosing Day 58 for Cycle 3.
Time Frame: as for outcome 11
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
ng/mL
  Dosing Day 30: number analyzed (Participants) | 86
  Dosing Day 30 | 0.0001196 (384)
  Dosing Day 58: number analyzed (Participants) | 72
  Dosing Day 58 | 0 (0)

19. Secondary Outcome: Clearance (CL) of Serum Inotuzumab Ozogamicin in Participants Receiving Inotuzumab+Rituximab on Dosing Day 30 and Day 58
Description: Clearance is defined as Dose/AUCinf. Study Days Cycle 2, Days 30 (0, 1, 4 hours), 32, 36, 38, 43, 50, and 57 and Cycle 3, Days 58 (0, 1, 4 hours), 60, 64, 66, 71, 78, and 85 correspond to Dosing Day 30 for Cycle 2 and Dosing Day 58 for Cycle 3.
Time Frame: as for outcome 11
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
L/hr
  Cycle 2 Day 30: number analyzed (Participants) | 32
  Cycle 2 Day 30 | 0.09855 (33)
  Cycle 3 Day 58: number analyzed (Participants) | 36
  Cycle 3 Day 58 | 0.08743 (37)

20. Secondary Outcome: Steady-state Volume of Distribution (Vss) of Inotuzumab Ozogamicin in Serum in Participants Receiving Inotuzumab MTD+Rituximab 375 mg/m^2 on Dosing Day 30 and Day 58
Description: Vss of inotuzumab ozogamicin on Dosing Days 30 and 58 were reported. Vss=CL*MRT (mean residence time). Study Days Cycle 2, Days 30 (0, 1, 4 hours), 32, 36, 38, 43, 50, and 57 and Cycle 3, Days 58 (0, 1, 4 hours), 60, 64, 66, 71, 78, and 85 correspond to Dosing Day 30 for Cycle 2 and Dosing Day 58 for Cycle 3.
Time Frame: as for outcome 11
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
L
  Dosing Day 30: number analyzed (Participants) | 32
  Dosing Day 30 | 4.860 (37)
  Dosing Day 58: number analyzed (Participants) | 36
  Dosing Day 58 | 5.183 (38)

21. Secondary Outcome: MRT of Inotuzumab Ozogamicin in Serum in Participants Receiving Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 on Dosing Day 30 and Day 58
Description: MRT: AUMCinf/AUCinf - DOF (degrees of freedom)/2, where AUMCinf is the area under the first moment curve derived using the linear/log trapezoidal method, and DOF is the duration of the IV infusion dose. Study Days Cycle 2, Days 30 (0, 1, 4 hours), 32, 36, 38, 43, 50, and 57 and Cycle 3, Days 58 (0, 1, 4 hours), 60, 64, 66, 71, 78, and 85 correspond to Dosing Day 30 for Cycle 2 and Dosing Day 58 for Cycle 3.
Time Frame: as for outcome 11
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
hr
  Dosing Day 30: number analyzed (Participants) | 32
  Dosing Day 30 | 49.31 (39)
  Dosing Day 58: number analyzed (Participants) | 36
  Dosing Day 58 | 59.24 (27)

22. Secondary Outcome: Serum Decay Half-Life (t1/2) of Inotuzumab Ozogamicin in Participants Receiving Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 on Dosing Day 30 and Day 58
Description: Termnial half-life (t½): Loge(2)/kel, where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
  Study Days Cycle 2, Days 30 (0, 1, 4 hours), 32, 36, 38, 43, 50, and 57 and Cycle 3, Days 58 (0, 1, 4 hours), 60, 64, 66, 71, 78, and 85 correspond to Dosing Day 30 for Cycle 2 and Dosing Day 58 for Cycle 3.
Time Frame: as for outcome 11
Population: PK population
Measure: Median (Full Range); unit: hr
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
hr
  Dosing Day 30: number analyzed (Participants) | 32
  Dosing Day 30 | 40.15 [15.4 to 78.4]
  Dosing Day 58: number analyzed (Participants) | 36
  Dosing Day 58 | 43.00 [30.5 to 57.6]

23. Secondary Outcome: AUCinf of Total Calicheamicin (Conjugated + Unconjugated) in Participants Receiving Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 on Dosing Day 30 and Day 58
Description: AUCinf: AUClast+(Clast/kel) where Clast is the predicted serum concentration at the last quantifiable timepoint estimated from the log-linear regression analysis. Study Days Cycle 2, Days 30 (0, 1, 4 hours), 32, 36, 38, 43, 50, and 57 and Cycle 3, Days 58 (0, 1, 4 hours), 60, 64, 66, 71, 78, and 85 correspond to Dosing Day 30 for Cycle 2 and Dosing Day 58 for Cycle 3.
Time Frame: as for outcome 11
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·hr/mL
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
ng·hr/mL
  Dosing Day 30: number analyzed (Participants) | 44
  Dosing Day 30 | 8437 (39)
  Dosing Day 58: number analyzed (Participants) | 37
  Dosing Day 58 | 10060 (58)

24. Secondary Outcome: AUClast of Total Calicheamicin (Conjugated Plus Unconjugated) in Participants Receiving Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 on Dosing Day 1, Day 30 and Day 58
Description: AUClast: AUC over dosage interval through last measurable time point, Tlast, using Linear/Log trapezoidal method. Study Days Cycle 1, Days 1 (0 hour), 2 (0, 1, 4 hours), 4, 8, 10, 15, and 29; Cycle 2, Days 30 (0, 1, 4 hours), 32, 36, 38, 43, 50, and 57; and Cycle 3, Days 58 (0, 1, 4 hours), 60, 64, 66, 71, 78, and 85 correspond to Dosing Day 1 for Cycle 1; Dosing Day 30 for Cycle 2; and Dosing Day 58 for Cycle 3.
Time Frame: as for outcome 12
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: n*hr/mL
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
n*hr/mL
  Dosing Day 1: number analyzed (Participants) | 100
  Dosing Day 1 | 1901 (192)
  Dosing Day 30: number analyzed (Participants) | 87
  Dosing Day 30 | 6129 (85)
  Dosing Day 58: number analyzed (Participants) | 71
  Dosing Day 58 | 6755 (145)

25. Secondary Outcome: Time of the Last Quantifiable Concentration in a Dosing Interval (Tlast) of Total Calicheamicin (Conjugated Plus Unconjugated) in Participants Receiving Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 on Dosing Day 1, Day 30 and Day 58
Description: Tlast: Time of last quantifiable concentration. Observed directly from data. Study Days Cycle 1, Days 1 (0 hour), 2 (0, 1, 4 hours), 4, 8, 10, 15, and 29; Cycle 2, Days 30 (0, 1, 4 hours), 32, 36, 38, 43, 50, and 57; and Cycle 3, Days 58 (0, 1, 4 hours), 60, 64, 66, 71, 78, and 85 correspond to Dosing Day 1 for Cycle 1; Dosing Day 30 for Cycle 2; and Dosing Day 58 for Cycle 3.
Time Frame: as for outcome 12
Population: PK population
Measure: Median (Full Range); unit: hr
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
hr
  Dosing Day 1: number analyzed (Participants) | 100
  Dosing Day 1 | 149 [1.25 to 647]
  Dosing Day 30: number analyzed (Participants) | 87
  Dosing Day 30 | 312 [4.17 to 654]
  Dosing Day 58: number analyzed (Participants) | 71
  Dosing Day 58 | 458 [1.00 to 650]

26. Secondary Outcome: Area Under the Steady-state Serum Concentration-time Curve (AUCtau) for Total Calicheamicin (Conjugated Plus Unconjugated) in Participants Receiving Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 on Dosing Day 1, Day 30, and Day 58
Description: AUCtau=AUC over dosage interval tau calculated using Linear/log trapezoidal method. Study Days Cycle 1, Days 1 (0 hour), 2 (0, 1, 4 hours), 4, 8, 10, 15, and 29; Cycle 2, Days 30 (0, 1, 4 hours), 32, 36, 38, 43, 50, and 57; and Cycle 3, Days 58 (0, 1, 4 hours), 60, 64, 66, 71, 78, and 85 correspond to Dosing Day 1 for Cycle 1; Dosing Day 30 for Cycle 2; and Dosing Day 58 for Cycle 3.
Time Frame: as for outcome 12
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·hr/mL
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
ng·hr/mL
  Dosing Day 1: number analyzed (Participants) | 39
  Dosing Day 1 | 3201 (78)
  Dosing Day 30: number analyzed (Participants) | 44
  Dosing Day 30 | 7794 (38)
  Dosing Day 58: number analyzed (Participants) | 37
  Dosing Day 58 | 9197 (54)

27. Secondary Outcome: Peak Serum Concentration (Cmax) of Total Calicheamicin (Conjugated Plus Unconjugated) in Participants Receiving Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 on Dosing Day 1, Day 30 and Day 58
Description: Cmax: Observed directly from data Study Days Cycle 1, Days 1 (0 hour), 2 (0, 1, 4 hours), 4, 8, 10, 15, and 29; Cycle 2, Days 30 (0, 1, 4 hours), 32, 36, 38, 43, 50, and 57; and Cycle 3, Days 58 (0, 1, 4 hours), 60, 64, 66, 71, 78, and 85 correspond to Dosing Day 1 for Cycle 1; Dosing Day 30 for Cycle 2; and Dosing Day 58 for Cycle 3.
Time Frame: as for outcome 12
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
ng/mL
  Dosing Day 1: number analyzed (Participants) | 103
  Dosing Day 1 | 54.36 (226)
  Dosing Day 30: number analyzed (Participants) | 89
  Dosing Day 30 | 58.67 (283)
  Dosing Day 58: number analyzed (Participants) | 73
  Dosing Day 58 | 64.43 (47)

28. Secondary Outcome: Time of Observed Maximum Concentration (Tmax) of Total Calicheamicin (Conjugated+Unconjugated) in Participants Receiving Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 on Dosing Day 1, Day 30 and Day 58
Description: as for outcome 16
Time Frame: as for outcome 12
Population: PK population
Measure: Median (Full Range); unit: hr
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
hr
  Dosing Day 1: number analyzed (Participants) | 102
  Dosing Day 1 | 1.05 [0 to 47.5]
  Dosing Day 30: number analyzed (Participants) | 88
  Dosing Day 30 | 1.26 [0.583 to 190]
  Dosing Day 58: number analyzed (Participants) | 73
  Dosing Day 58 | 1.38 [0 to 478]

29. Secondary Outcome: Average Serum Concentration (Cav) of Total Calicheamicin (Conjugated Plus Unconjugated) in Participants Receiving Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 on Dosing Day 30 and Day 58
Description: Cav: AUCtau/tau for Dosing Day 30 Cycle 2 and Dosing Day 58 Cycle 3. Study Days Cycle 2, Days 30 (0, 1, 4 hours), 32, 36, 38, 43, 50, and 57 and Cycle 3, Days 58 (0, 1, 4 hours), 60, 64, 66, 71, 78, and 85 correspond to Dosing Day 30 for Cycle 2 and Dosing Day 58 for Cycle 3.
Time Frame: as for outcome 11
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
ng/mL
  Dosing Day 30: number analyzed (Participants) | 44
  Dosing Day 30 | 11.60 (38)
  Dosing Day 58: number analyzed (Participants) | 37
  Dosing Day 58 | 13.69 (54)

30. Secondary Outcome: Minimum Observed Serum Trough Concentration (Cmin) of Total Calicheamicin (Conjugated Plus Unconjugated) in Participants Receiving Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 on Dosing Day 30 and Day 58
Description: Cmin: Lowest concentration observed during the dosing interval tau. Observed directly from data from Day 30 for Cycle 2; and Day 58 for Cycle 3. Study Days Cycle 2, Days 30 (0, 1, 4 hours), 32, 36, 38, 43, 50, and 57 and Cycle 3, Days 58 (0, 1, 4 hours), 60, 64, 66, 71, 78, and 85 correspond to Dosing Day 30 for Cycle 2 and Dosing Day 58 for Cycle 3.
Time Frame: as for outcome 11
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
ng/mL
  Dosing Day 30: number analyzed (Participants) | 88
  Dosing Day 30 | 0.0001326 (564)
  Dosing Day 58: number analyzed (Participants) | 73
  Dosing Day 58 | 0.0001350 (497)

31. Secondary Outcome: Clearance (CL) of Total Calicheamicin (Conjugated Plus Unconjugated) in Participants Receiving Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 on Dosing Day 30 and Day 58
Description: Clearance defined as Dose/AUCinf. Corresponds to Dosing Day 30 for Cycle 2 and dosing Day 58 for Cycle 3. Study Days Cycle 2, Days 30 (0, 1, 4 hours), 32, 36, 38, 43, 50, and 57 and Cycle 3, Days 58 (0, 1, 4 hours), 60, 64, 66, 71, 78, and 85 correspond to Dosing Day 30 for Cycle 2 and Dosing Day 58 for Cycle 3.
Time Frame: as for outcome 11
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
L/hr
  Dosing Day 30: number analyzed (Participants) | 44
  Dosing Day 30 | 0.4353 (40)
  Dosing Day 58: number analyzed (Participants) | 37
  Dosing Day 58 | 0.3799 (57)

32. Secondary Outcome: Steady-state Volume (Vss) of Total Calicheamicin (Conjugated Plus Unconjugated) Distribution in Participants Receiving Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 on Dosing Day 30 and Day 58
Description: Vss: Steady-state volume of distribution CL*MRT of inotuzumab ozogamicin Day 30 for Cycle 2; and Day 58 for Cycle 3. Study Days Cycle 2, Days 30 (0, 1, 4 hours), 32, 36, 38, 43, 50, and 57 and Cycle 3, Days 58 (0, 1, 4 hours), 60, 64, 66, 71, 78, and 85 correspond to Dosing Day 30 for Cycle 2 and Dosing Day 58 for Cycle 3.
Time Frame: as for outcome 11
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
L
  Dosing Day 30: number analyzed (Participants) | 44
  Dosing Day 30 | 72.95 (35)
  Dosing Day 58: number analyzed (Participants) | 37
  Dosing Day 58 | 75.81 (26)

33. Secondary Outcome: Mean Residence Time (MRT) of Total Calicheamicin (Conjugated Plus Unconjugated) in Participants Receiving Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 on Dosing Day 30 and Day 58
Description: MRT: AUMCinf/AUCinf - DOF/2, where AUMCinf is the area under the first moment curve derived using the linear/log trapezoidal method, and DOF is the duration of the IV infusion dose. Study Days Cycle 2, Days 30 (0, 1, 4 hours), 32, 36, 38, 43, 50, and 57 and Cycle 3, Days 58 (0, 1, 4 hours), 60, 64, 66, 71, 78, and 85 correspond to Dosing Day 30 for Cycle 2 and Dosing Day 58 for Cycle 3.
Time Frame: as for outcome 11
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
hr
  Dosing Day 30: number analyzed (Participants) | 44
  Dosing Day 30 | 167.5 (41)
  Dosing Day 58: number analyzed (Participants) | 37
  Dosing Day 58 | 199.5 (49)

34. Secondary Outcome: Serum Decay Half-Life (t1/2) of Total Calicheamicin (Conjugated Plus Unconjugated) in Participants Receiving Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 on Dosing Day 30 and Day 58
Description: as for outcome 22
Time Frame: as for outcome 11
Population: Pk population
Measure: Median (Full Range); unit: hr
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
hr
  Dosing Day 30: number analyzed (Participants) | 44
  Dosing Day 30 | 126.5 [50.0 to 251]
  Dosing Day 58: number analyzed (Participants) | 37
  Dosing Day 58 | 176.0 [19.0 to 354]

35. Secondary Outcome: Area Under the Steady-state Serum Concentration-time Curve (AUClast) of Unconjugated Calicheamicin in Participants Receiving Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 on Dosing Day 1, Day 30 and Day 58
Description: as for outcome 24
Time Frame: as for outcome 12
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·hr/mL
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
ng·hr/mL
  Dosing Day 1: number analyzed (Participants) | 98
  Dosing Day 1 | 0.0009904 (22500000)
  Dosing Day 30: number analyzed (Participants) | 83
  Dosing Day 30 | 0.002008 (64300000)
  Dosing Day 58: number analyzed (Participants) | 68
  Dosing Day 58 | 0.005896 (1370000000)

36. Secondary Outcome: Time of the Last Quantifiable Concentration in a Dosing Interval (Tlast) of Unconjugated Calicheamicin in Participants Receiving Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 on Dosing Day 1, Day 30 and Day 58
Description: as for outcome 25
Time Frame: as for outcome 12
Population: PK population
Measure: Median (Full Range); unit: hr
Groups:
- INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2: Participants received the MTD determined in the dose escalation phase; MTD determination in the dose escalation phase was based on toxicities during the first cycle. Participants with follicular lymphoma, DLBCL, and refractory aggressive or intermediate B-cell NHL received rituximab 375 mg/m^2 via IV infusion on Day 1 and the MTD of inotuzumab ozogamicin (1.8 mg/m^2) via IV infusion on Day 2 of each 28-day cycle for up to 8 cycles unless there was evidence of progressive disease, unacceptable toxicity, or the participant refused further treatment.
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
hr
  Dosing Day 1: number analyzed (Participants) | 18
  Dosing Day 1 | 48.5 [1.00 to 674]
  Dosing Day 30: number analyzed (Participants) | 22
  Dosing Day 30 | 4.00 [1.00 to 648]
  Dosing Day 58: number analyzed (Participants) | 26
  Dosing Day 58 | 4.00 [0 to 1060]

37. Secondary Outcome: Peak Serum Concentration (Cmax) of Unconjugated Calicheamicin in Participants Receiving Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 on Dosing Day 1, Day 30 and Day 58
Description: as for outcome 27
Time Frame: as for outcome 12
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
ng/mL
  Dosing Day 1: number analyzed (Participants) | 103
  Dosing Day 1 | 0.0005608 (121496)
  Dosing Day 30: number analyzed (Participants) | 89
  Dosing Day 30 | 0.001153 (1020000)
  Dosing Day 58: number analyzed (Participants) | 73
  Dosing Day 58 | 0.003250 (6780000)

38. Secondary Outcome: Time of Observed Maximum Concentration (Tmax) of Unconjugated Calicheamicin in Participants Receiving Inotuzumab Ozogamicin + Rituximab on Dosing Day 1, Day 30 and Day 58
Description: as for outcome 16
Time Frame: as for outcome 12
Population: PK population
Measure: Median (Full Range); unit: hr
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
hr
  Dosing Day 1: number analyzed (Participants) | 18
  Dosing Day 1 | 1.38 [0.983 to 647]
  Dosing Day 30: number analyzed (Participants) | 22
  Dosing Day 30 | 4.00 [1.00 to 47.0]
  Dosing Day 58: number analyzed (Participants) | 26
  Dosing Day 58 | 3.42 [0 to 1060]

39. Secondary Outcome: Minimum Observed Serum Trough Concentration (Cmin) of Unconjugated Calicheamicin in Participants Receiving Inotuzumab Ozogamicin+Rituximab on Dosing Day 30 and Day 58
Description: Cmin: Lowest concentration observed during the dosing interval tau. Study Days Cycle 2, Days 30 (0, 1, 4 hours), 32, 36, 38, 43, 50, and 57 and Cycle 3, Days 58 (0, 1, 4 hours), 60, 64, 66, 71, 78, and 85 correspond to Dosing Day 30 for Cycle 2 and Dosing Day 58 for Cycle 3.
Time Frame: as for outcome 11
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
ng/mL
  Dosing Day 30: number analyzed (Participants) | 22
  Dosing Day 30 | 0.0001588 (1044)
  Dosing Day 58: number analyzed (Participants) | 26
  Dosing Day 58 | 0.0001495 (811)

40. Secondary Outcome: Area Under the Serum Concentration-time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) of Inotuzumab Ozogamicin Antibody in Participants Receiving Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m2 on Dosing Day 30 and Day 58
Description: as for outcome 23
Time Frame: as for outcome 11
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·hr/mL
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
ng·hr/mL
  Dosing Day 30: number analyzed (Participants) | 68
  Dosing Day 30 | 83270 (36)
  Dosing Day 58: number analyzed (Participants) | 60
  Dosing Day 58 | 93760 (30)

41. Secondary Outcome: Area Under the Steady-state Concentration-time Curve (AUClast) of Serum Inotuzumab Ozogamicin Antibody in Participants Receiving Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 on Dosing Day 1, Day 30 and Day 58
Description: as for outcome 24
Time Frame: as for outcome 12
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·hr/mL
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
ng·hr/mL
  Dosing Day 1: number analyzed (Participants) | 100
  Dosing Day 1 | 25740 (139)
  Dosing Day 30: number analyzed (Participants) | 87
  Dosing Day 30 | 61770 (88)
  Dosing Day 58: number analyzed (Participants) | 71
  Dosing Day 58 | 72430 (95)

42. Secondary Outcome: Time of the Last Quantifiable Concentration in a Dosing Interval (Tlast) of Serum Inotuzumab Ozogamicin Antibody in Participants Receiving Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 on Dosing Day 1, Day 30 and Day 58
Description: as for outcome 25
Time Frame: as for outcome 12
Population: PK population
Measure: Median (Full Range); unit: hr
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
hr
  Dosing Day 1: number analyzed (Participants) | 100
  Dosing Day 1 | 190 [1.25 to 502]
  Dosing Day 30: number analyzed (Participants) | 87
  Dosing Day 30 | 310 [4.00 to 505]
  Dosing Day 58: number analyzed (Participants) | 71
  Dosing Day 58 | 312 [3.58 to 648]

43. Secondary Outcome: Serum Decay Half-Life (t1/2) of Inotuzumab Ozogamicin Antibody in Participants Receiving Inotuzumab Ozogamicin MTD + Rituximab on Dosing Day 30 and Day 58
Description: as for outcome 22
Time Frame: as for outcome 11
Population: PK population
Measure: Median (Full Range); unit: hr
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
hr
  Dosing Day 30: number analyzed (Participants) | 68
  Dosing Day 30 | 99.35 [37.8 to 153]
  Dosing Day 58: number analyzed (Participants) | 60
  Dosing Day 58 | 103.5 [58.6 to 172]

44. Secondary Outcome: Area Under the Steady-state Serum Concentration-time Curve (AUCtau) of Inotuzumab Ozogamicin Antibody in Participants Receiving Inotuzumab Ozogamicin MTD+ Rituximab 375 mg/m^2 on Dosing Day 1, Day 30, and Day 58
Description: as for outcome 26
Time Frame: as for outcome 12
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·hr/mL
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
ng·hr/mL
  Dosing Day 1: number analyzed (Participants) | 75
  Dosing Day 1 | 40180 (51)
  Dosing Day 30: number analyzed (Participants) | 68
  Dosing Day 30 | 80060 (37)
  Dosing Day 58: number analyzed (Participants) | 60
  Dosing Day 58 | 91370 (32)

45. Secondary Outcome: Peak Concentration (Cmax) of Serum Inotuzumab Ozogamicin Antibody in Participants Receiving Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 on Dosing Day 1, Day 30 and Day 58
Description: as for outcome 27
Time Frame: as for outcome 12
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
ng/mL
  Dosing Day 1: number analyzed (Participants) | 101
  Dosing Day 1 | 776.6 (36)
  Dosing Day 30: number analyzed (Participants) | 89
  Dosing Day 30 | 700.4 (448)
  Dosing Day 58: number analyzed (Participants) | 73
  Dosing Day 58 | 653.0 (625)

46. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) of Serum Inotuzumab Ozogamicin Antibody in Participants Receiving Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 on Dosing Day 1, Day 30 and Day 58
Description: as for outcome 16
Time Frame: as for outcome 12
Population: PK population
Measure: Median (Full Range); unit: hr
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
hr
  Dosing Day 1: number analyzed (Participants) | 101
  Dosing Day 1 | 1.05 [0 to 6.58]
  Dosing Day 30: number analyzed (Participants) | 88
  Dosing Day 30 | 1.17 [0.700 to 146]
  Dosing Day 58: number analyzed (Participants) | 72
  Dosing Day 58 | 3.79 [0 to 478]

47. Secondary Outcome: Average Serum Concentration (Cav) of Inotuzumab Ozogamicin Antibody in Participants Receiving Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 on Dosing Day 30 and Day 58
Description: as for outcome 29
Time Frame: as for outcome 11
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
ng/mL
  Dosing Day 30: number analyzed (Participants) | 68
  Dosing Day 30 | 119.2 (37)
  Dosing Day 58: number analyzed (Participants) | 60
  Dosing Day 58 | 136 (32)

48. Secondary Outcome: Minimum Observed Serum Trough Concentration (Cmin) of Inotuzumab Ozogamicin Antibody in Participants Receiving Inotuzumab MTD + Rituximab 375 mg/m^2 on Dosing Day 30 and Day 58
Description: as for outcome 39
Time Frame: as for outcome 11
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
ng/mL
  Dosing Day 30: number analyzed (Participants) | 88
  Dosing Day 30 | 0.0001190 (366)
  Dosing Day 58: number analyzed (Participants) | 72
  Dosing Day 58 | 0 (0)

49. Secondary Outcome: Clearance (CL) of Serum Inotuzumab Ozogamicin Antibody in Participants Receiving Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 on Dosing Day 30 and Day 58
Description: Clearance defined as Dose/AUCinf. Study Days Cycle 2, Days 30 (0, 1, 4 hours), 32, 36, 38, 43, 50, and 57 and Cycle 3, Days 58 (0, 1, 4 hours), 60, 64, 66, 71, 78, and 85 correspond to Dosing Day 30 for Cycle 2 and Dosing Day 58 for Cycle 3.
Time Frame: as for outcome 11
Population: PK populatoin
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
L/hr
  Dosing Day 30: number analyzed (Participants) | 68
  Dosing Day 30 | 0.04240 (41)
  Dosing Day 58: number analyzed (Participants) | 60
  Dosing Day 58 | 0.03699 (36)

50. Secondary Outcome: Steady-state Volume (Vss) of Inotuzumab Ozogamicin Antibody Distribution in Participants Receiving Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 on Dosing Day 30 and Day 58
Description: as for outcome 32
Time Frame: as for outcome 11
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Groups:
- INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2: Participants received the MTD determined in the dose escalation phase; MTD determination in the dose escalation phase was based on toxicities during the 1st cycle. Participants with follicular lymphoma, DLBCL, and refractory aggressive or intermediate B-cell NHL received rituximab 375 mg/m^2 via IV infusion on Day 1 and the MTD of inotuzumab ozogamicin (1.8 mg/m^2) via IV infusion on Day 2 of each 28-day cycle for up to 8 cycles unless there was evidence of progressive disease, unacceptable toxicity, or the participant refused further treatment.
Arm/Group | INOTUZUMAB OZOGAMICIN MTD + RITUXIMAB 375 MG/M^2
Number analyzed (Participants) | 104
L
  Dosing Day 30: number analyzed (Participants) | 68
  Dosing Day 30 | 5.283 (29)
  Dosing Day 58: number analyzed (Participants) | 60
  Dosing Day 58 | 4.952 (34)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded and reported from the time a participant signed the Informed Consent Form (ICF) until at least 28 days after last dose of study treatment. Summarized data reflects incidents from 1st dose to up to 56 days post last dose.
Description: The same event may appear as both an AE and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another participant, or 1 participant may have experienced both a serious and nonserious event during the study.
Groups:
- Inotuzumab Ozogamicin 0.8 mg/m^2+ Rituximab 375 mg/m^2: Participants received rituximab 375 mg/m^2 via IV infusion on Day 1 and inotuzumab ozogamicin 0.8 mg/m^2 via IV infusion on Day 2 of each 28-day cycle for up to 8 cycles unless there was evidence of progressive disease, unacceptable toxicity, or the subject refused further treatment.
- Inotuzumab Ozogamicin 1.3 mg/m^2+ Rituximab 375 mg/m^2: Participants received rituximab 375 mg/m^2 via IV infusion on Day 1 and inotuzumab ozogamicin 1.3 mg/m^2 via IV infusion on Day 2 of each 28-day cycle for up to 8 cycles unless there was evidence of progressive disease, unacceptable toxicity, or the subject refused further treatment.
- Inotuzumab Ozogamicin 1.8 mg/m^2+ Rituximab 375 mg/m^2: Participants received rituximab 375 mg/m^2 via IV infusion on Day 1 and inotuzumab ozogamicin 1.8 mg/m^2 via IV infusion on Day 2 of each 28-day cycle for up to 8 cycles unless there was evidence of progressive disease, unacceptable toxicity, or the subject refused further treatment.
- Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 Follicular: Participants received the MTD determined in the dose escalation phase; MTD determination in the dose escalation phase was based on toxicities during the 1st cycle. Participants with follicular lymphoma received rituximab 375 mg/m^2 via IV infusion on Day 1 and the MTD of inotuzumab ozogamicin (1.8 mg/m^2) via IV infusion on Day 2 of each 28-day cycle for up to 8 cycles unless there was evidence of progressive disease, unacceptable toxicity, or the subject refused further treatment.
- Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 DLBCL: Participants received the MTD determined in the dose escalation phase; MTD determination in the dose escalation phase was based on toxicities during the 1st cycle. Participants with DLBCL received rituximab 375 mg/m^2 via IV infusion on Day 1 and the MTD of inotuzumab ozogamicin (1.8 mg/m^2) via IV infusion on Day 2 of each 28-day cycle for up to 8 cycles unless there was evidence of progressive disease, unacceptable toxicity, or the subject refused further treatment.
- Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 Refractory: Participants received the MTD determined in the dose escalation phase; MTD determination in the dose escalation phase was based on toxicities during the 1st cycle. Participants with either refractory aggressive or intermediate B-cell NHL received rituximab 375 mg/m^2 via IV infusion on Day 1 and the MTD of inotuzumab ozogamicin (1.8 mg/m^2) via IV infusion on Day 2 of each 28-day cycle for up to 8 cycles unless there was evidence of progressive disease, unacceptable toxicity, or the subject refused further treatment.
Arm/Group | Inotuzumab Ozogamicin 0.8 mg/m^2+ Rituximab 375 mg/m^2 | Inotuzumab Ozogamicin 1.3 mg/m^2+ Rituximab 375 mg/m^2 | Inotuzumab Ozogamicin 1.8 mg/m^2+ Rituximab 375 mg/m^2 | Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 Follicular | Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 DLBCL | Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 Refractory
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/3 | 1/7 | 9/34 | 12/40 | 5/30
Other Adverse Events (participants affected / at risk) | 5/5 | 3/3 | 7/7 | 34/34 | 39/40 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inotuzumab Ozogamicin 0.8 mg/m^2+ Rituximab 375 mg/m^2 (N=5) | Inotuzumab Ozogamicin 1.3 mg/m^2+ Rituximab 375 mg/m^2 (N=3) | Inotuzumab Ozogamicin 1.8 mg/m^2+ Rituximab 375 mg/m^2 (N=7) | Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 Follicular (N=34) | Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 DLBCL (N=40) | Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 Refractory (N=30)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Shock (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Visceroptosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Disease progression (General disorders) | 1 | 0 | 0 | 0 | 1 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Local swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bundle branch block left (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Candida pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Intervertebral discitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Pneumonia klebsiella (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Spider naevus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Inotuzumab Ozogamicin 0.8 mg/m^2+ Rituximab 375 mg/m^2 (N=5) | Inotuzumab Ozogamicin 1.3 mg/m^2+ Rituximab 375 mg/m^2 (N=3) | Inotuzumab Ozogamicin 1.8 mg/m^2+ Rituximab 375 mg/m^2 (N=7) | Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 Follicular (N=34) | Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 DLBCL (N=40) | Inotuzumab Ozogamicin MTD + Rituximab 375 mg/m^2 Refractory (N=30)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 3 | 7 | 3
Hyperfibrinogenaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 5 | 5 | 4
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1 | 9 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 4 | 18 | 11 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2 | 5 | 15 | 27 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 5 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 4 | 5 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 3 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 3 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 6 | 4 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 2 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 1 | 1 | 0 | 3 | 3 | 1
Hot flush (Vascular disorders) | 1 | 0 | 0 | 3 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 3 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1 | 2 | 1 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 4 | 5 | 1
Eye pain (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 4 | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 4 | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 6 | 4 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 3 | 1 | 2
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 3
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 9 | 13 | 5
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 9 | 8 | 9
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 5 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 3 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 5 | 24 | 24 | 11
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2 | 0
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 3 | 13 | 8 | 7
Asthenia (General disorders) | 1 | 0 | 1 | 2 | 4 | 1
Catheter site erythema (General disorders) | 0 | 1 | 0 | 0 | 1 | 0
Catheter site pruritus (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 2 | 1 | 2 | 1
Chest pain (General disorders) | 0 | 0 | 1 | 1 | 0 | 0
Chills (General disorders) | 1 | 1 | 2 | 4 | 12 | 2
Crepitations (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 5 | 1 | 5 | 16 | 22 | 13
Influenza like illness (General disorders) | 0 | 0 | 1 | 4 | 0 | 1
Local swelling (General disorders) | 0 | 0 | 1 | 0 | 2 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Oedema (General disorders) | 0 | 0 | 0 | 2 | 2 | 0
Oedema peripheral (General disorders) | 1 | 1 | 1 | 4 | 7 | 4
Pain (General disorders) | 0 | 0 | 1 | 1 | 1 | 2
Pyrexia (General disorders) | 0 | 1 | 4 | 12 | 8 | 7
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 2
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 2 | 2 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 2
Oropharyngitis fungal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 3 | 3 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 5 | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 4 | 5 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 3 | 5 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 9 | 11 | 9
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 3 | 17 | 18 | 10
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 2 | 15 | 13 | 7
Blood bilirubin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2
Blood cholesterol increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 2
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 1 | 2 | 3
Blood fibrinogen increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 2 | 9 | 13 | 6
Blood triglycerides increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood urea increased (Investigations) | 1 | 0 | 0 | 0 | 3 | 1
Blood urine present (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 3
Fibrin D dimer increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 1 | 4 | 3
Monocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2
Protein total increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 2
Urine protein/creatinine ratio increased (Investigations) | 0 | 0 | 0 | 0 | 3 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 3 | 6 | 5
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 2 | 1 | 2
Urine odour abnormal (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 12 | 13 | 9
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 2 | 9 | 6 | 6
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 7 | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 5 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 5 | 6 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 7 | 2 | 1
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 3 | 3
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 11 | 6 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 3 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 3 | 12 | 5 | 5
Hypogeusia (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 7 | 3 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 2 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 2 | 2 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 1 | 2 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 3 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 4 | 4 | 1
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 0 | 0
Nipple pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 9 | 5 | 8
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 9 | 6 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 9 | 8 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 5 | 1 | 3
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 1 | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 4 | 1 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 2 | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 6 | 3 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No